CLINICAL TRIAL: NCT05817058
Title: A Phase 1 Multicenter, Open Label, First-in-Human Dose Escalation Study of AFM28, a Bispecific ICE® That Targets CD123 and CD16A, in Patients With CD123-Positive Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: First-in-Human Dose Escalation Study of AFM28 in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: As decided by sponsor
Sponsor: Affimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFM28-101
Record Dates: First submitted 2023-03-22; First posted 2023-04-18 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of escalating doses of AFM28 (Experimental): AFM28 first in human starting dose will be 25 mg i.v.
  Interventions: Drug: AFM28

INTERVENTIONS:
Drug: AFM28 — AFM28 dose escalation

SUMMARY:
This study is a First In Human, phase 1, open-label, non-randomized, multi-center, multiple ascending dose escalation study evaluating AFM28 as a monotherapy in subjects with Relapsed/Refractory CD123-positive Acute Myeloid Leukemia (AML). AFM28 is a tetravalent monoclonal antibody targeting the interleukin-3 receptor subunit alpha (IL3RA, CD123) and the low affinity immunoglobulin gamma Fc region receptor III-A (FCGR3A, CD16A). It is developed as an antineoplastic agent for hematologic malignancies known to express CD123. The primary pharmacological Mode of Action of AFM28 is induction of cell death of CD123-expressing cells by stimulating Antibody-Dependent Cell-mediated Cytotoxicity mediated by CD16A-expressing immune cells, primarily Natural Killer cells. The aim of the dose escalation is to determine the Maximum Tolerated Dose (MTD) and/or establish one or more Recommended Phase 2 Doses, based on safety, preliminary anti-leukemic activity and Pharmacokinetics / Pharmacodynamics data.

DETAILED DESCRIPTION:
The study drug will be given by intravenous infusion once weekly as long as the subject is deriving clinical benefit until disease progression or other treatment discontinuation criteria met, unacceptable toxicity, or subject's refusal, whichever occurs first. The dose-limiting toxicity observation period will be 28 days, reflecting adequate exposure for safety assessment. The dose-escalation scheme will follow a Bayesian logistic regression model. A safety review committee will monitor safety and recommend all cohort dosing decisions. The starting First In Human dose for AFM28 will be 25 mg i.v. and treatment in each cohort will utilize a staggered approach, with at least 7 days between the first dose of the first subject and the first dose of subsequent subjects. In order to gather additional Pharmacokinetics/ Pharmacodynamics and safety data to inform potential final dose escalation decisions and selection of one or more recommended phase 2 doses at selected dose levels, additional subjects may be enrolled in at least two cohorts consistent with backfilling a cohort (up to 12 subjects).

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects with a confirmed diagnosis of AML as defined by 2016 WHO Classification and determined by pathology review at the study site. Subjects with acute promyelocytic leukemia are excluded.

  2. Subjects must have CD123-positive AML confirmed on bone marrow or peripheral blood at Screening (assessed locally without any cut-off level).

  3. Subjects with AML who are in the first, second, or third relapse OR who are at least primary refractory and received at most 3 regimes of previous standard anti-leukemia therapy.

  4. Primary refractory is defined as ≥ 5% blasts in bone marrow following 2 cycles of anthracycline and cytarabine based induction (such as 3+7 or similar), or one cycle of purine analogue containing induction, or after ≥ 3 cycles hypomethylating agent ± or low dose cytarabine ± B-Cell lymphoma 2 based induction regimen, or ≥ 4 cycles of hypomethylating agent based therapy.

  5. Subjects with prior autologous and allogeneic bone marrow transplant are eligible. Subjects with an allogeneic transplant must meet the following conditions: The transplant must have been performed > 3 months before the date of dosing on this study, the subject must not have active graft versus host disease, must be off all graft versus host disease medications at least > 28 days prior to date of dosing of study drug (for example, calcineurin inhibitors, ≥ 10 mg/day prednisone or other steroid equivalent, or other immunosuppressive agents).

Exclusion Criteria:

* 1. Diagnosis of BCR-ABL-positive leukemia, acute promyelocytic leukemia, or juvenile myelomonocytic leukemia.

  2. Known hypersensitivity/allergic reaction ≥ grade 3 to monoclonal antibodies or any components used in the AFM28 drug product preparation, any history of anaphylaxis or uncontrolled asthma. Prior CD123 targeting therapies should be allowed after discussion with and at the discretion of the Sponsor.

  3. Received any anticancer therapy or investigational treatment for AML within 14 days of the first dose of study drug and within 28 days for biological agents including but not limited to monoclonal antibodies, cellular therapies, bispecific antibodies, checkpoint antibodies and others. Must have recovered to grade ≤ 1 from any grade 2 to 4 toxicity from previous treatment, except alopecia.

  4. History of any other systemic malignancy, unless previously treated with curative intent and the subject has been disease free for 2 years or longer. Examples for acceptable previous malignancies include completely removed in situ cervical intra-epithelial neoplasia, non-melanoma skin cancer, ductal carcinoma in situ, early-stage prostate cancer that has been adequately treated. Subjects who meet the above criteria and are on maintenance therapy for the prior malignancy may be eligible after discussion and approval from the medical monitor.

  5. The subject has received radionuclide treatment within 6 weeks of the first dose of study treatment.

  6. Known clinically active or suspected central nervous system (CNS) leukemia. If suspected, CNS leukemia should be ruled out with relevant imaging and/or examination of cerebrospinal fluid. Subjects with known prior CNS leukemia should have had at least two consecutive negative Lumbar Punctures for CNS leukemia and no clinical signs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
The Incidence of dose limiting toxicities | 28 days following the first dose of study treatment
  The incidence of dose limiting toxicities during dose limiting toxicities observation period considering the totality of treatment-emergent adverse events is evaluated using
  * National Cancer Institute Common Terminology Criteria for Adverse Events, v5.0
  * the American Society of Transplantation and Cellular Therapy Cytokine Release Syndrome grading system for Cytokine Release Syndrome
  * the Cairo-Bishop Tumor Lysing Syndrom (TLS) grading system for TLS

SECONDARY OUTCOMES:
Incidence and severity of Treatment Emergent Adverse Events | through study completion (up to 36 weeks)
  Incidence and severity of Treatment Emergent Adverse Events
Incidence and severity of Serious Adverse Events | through study completion (up to 36 weeks)
  Incidence and severity of Serious Adverse Events
Incidence of subjects developing anti-drug antibodies | through study completion (up to 36 weeks)
  Incidence of anti-drug antibodies during treatment with AFM28 (by measurement of anti-drug antibodies before and throughout treatment with AFM28)
Area under the concentration-time curve | cycle 1 (day 1 and day 28)
  Area under the concentration-time curve over the dose interval
Cmax | cycle 1 (day 1 and day 28)
  Maximum observed plasma concentration
Tmax | cycle 1 (day 1 and day 28)
  Time to reach maximum observed plasma concentration
Ctrough | immediately prior to the fourth dose
  Concentration measured immediately prior to the fourth dose
Complete Response | Through treatment period until 14 days after last dose
  Complete response (Disease assessment in accordance with the International Working Group (IWG) criteria for AML and the European Leukemia Network (ELN) 2017 classification criteria)
Complete Response hematological | Through treatment period until 14 days after last dose
  Complete Response with partial hematologic recovery (Disease assessment in accordance with the IWG criteria for AML and the ELN 2017 classification criteria)
Complete Response composite rate | Through treatment period until 14 days after last dose
  Composite complete response rate (Disease assessment in accordance with the IWG criteria for AML and the ELN 2017 classification criteria)
Complete Response + Complete Response hematological rate | Through treatment period until 14 days after last dose
  Complete Response plus Complete Response with partial hematologic recovery rate (Disease assessment in accordance with the IWG criteria for AML and the ELN 2017 classification criteria)
Overall Response Rate | Through treatment period until 14 days after last dose
  Overall response rate (Disease assessment in accordance with the IWG criteria for AML and the ELN 2017 classification criteria)
Disease Control Rate | Through treatment period until 14 days after last dose
  Disease control rate (Disease assessment in accordance with the IWG criteria for AML and the ELN 2017 classification criteria)
Duration of Response | Through treatment period until 14 days after last dose
  Duration of Response (Disease assessment in accordance with the IWG criteria for AML and the ELN 2017 classification criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Wunderle, Study Director — Affimed GmbH
Locations (5):
- France (2):
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Spain (3):
  - Institut Català d'Oncologia-Hospital Duran i Reynals, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No